CLINICAL TRIAL: NCT04855045
Title: An Open-Label, Dose Escalation and Double-Masked, Randomized, Controlled Study to Evaluate the Safety and Tolerability of Sepofarsen in Pediatric Subjects <8 Years of Age With Leber Congenital Amaurosis Type 10 (LCA10) Due to the c.2991 +1655A>G (p.Cys998X) Mutation.
Brief Title: An Open-label, Dose Escalation and Double-masked, Randomized, Controlled Trial Evaluating Safety and Tolerability of Sepofarsen in Children (<8 Years of Age) With LCA10 Caused by Mutations in the CEP290 Gene.
Acronym: BRIGHTEN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ProQR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PQ-110-005
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Leber Congenital Amaurosis 10; Blindness; Leber Congenital Amaurosis; Vision Disorders; Sensation Disorders; Neurologic Manifestations; Eye Diseases; Eye Disorders Congenital; Retinal Disease; Retinal Degeneration; Retinal Dystrophies
Keywords: LCA10; CEP290; p.Cys998X; c.2991+1655A>G; Leber Congenital Amaurosis; Antisense oligonucleotide; RNA therapy; QR-110; sepofarsen; pediatric; children
MeSH Terms: conditions — Leber Congenital Amaurosis 10; Blindness; Leber Congenital Amaurosis; Vision Disorders; Sensation Disorders; Neurologic Manifestations; Eye Diseases; Eye Abnormalities; Retinal Diseases; Retinal Degeneration; Retinal Dystrophies; Meckel Syndrome, Type 4

STUDY DESIGN:
Intervention Model Description: The study consists of two parts: an open-label dose escalation part, followed by a double-masked randomized part.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 - open label (Experimental)
  Interventions: Drug: sepofarsen
- Group 2 - open label (Experimental)
  Interventions: Drug: sepofarsen
- Group 3: open label (Experimental)
  Interventions: Drug: sepofarsen
- Group 4: double-masked, randomized to one of 2 dose cohorts (Experimental)
  Interventions: Drug: sepofarsen

INTERVENTIONS:
Drug: sepofarsen — RNA antisense oligonucleotide for intravitreal injection
  Other Names: QR-110

SUMMARY:
PQ-110-005 (BRIGHTEN) is an open-label, dose escalation and double-masked, randomized, controlled study evaluating safety and tolerability of sepofarsen administered via intravitreal (IVT) injection in pediatric subjects (<8 years of age) with LCA10 due to the c.2991+1655A>G mutation over 24 months of treatment.

DETAILED DESCRIPTION:
This is an open-label, dose escalation and double-masked, randomized, controlled study evaluating safety and tolerability of sepofarsen administered via intravitreal (IVT) injection in pediatric subjects (<8 years of age) with LCA10 due to the c.2991+1655A>G mutation. The study consists of two parts: an open-label dose escalation part, followed by a double-masked randomized part.

In the open label part; subjects will be assigned to one of 3 planned dose groups using a staggered dose escalation design. After at least 1 patient is dosed in each group; the Data Monitoring Committee (DMC) will review at least 4 weeks of safety data post dosing; and may recommend initiation of the next dose group. The DMC may recommend initiation of the double-masked randomized part of the study after completion of the last dose group in the dose escalation part of the study.

In the double-masked, randomized, controlled part of the study; subjects will be randomized to one of 2 planned dose groups .

Subjects will receive a unilateral IVT injection of sepofarsen on Day 1. Thereafter a 6-monthly dosing schedule is planned.

After each dosing subjects will be assessed for safety and tolerability at follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child, <8 years of age at Screening with a clinical diagnosis of LCA and a molecular diagnosis of homozygosity or compound heterozygosity for the CEP290 p.Cys998X mutation, based on genotyping analysis at Screening. A historic genotyping report from a certified laboratory are acceptable with Sponsor approval.
* BCVA equal to or better than Logarithm of the Minimum Angle of Resolution (logMAR) + 4.0 (Light Perception), and equal to or worse than logMAR + 0.4 in the treatment eye.
* Detectable outer nuclear layer (ONL) in the area of the macula.

Exclusion Criteria:

* Presence of any significant ocular or non-ocular disease/disorder which may put the subject at risk because of participation in the trial' may influence the results of the trial, or the subject's ability to participate in the trial.
* Receipt within 1 month prior to Screening of any intraocular or periocular surgery (including refractive surgery), or an IVT injection or planned intraocular surgery or procedure during the course of the trial.
* Current treatment or treatment within the past 12 months with therapies known to influence the immune system (including but not limited to cytostatics, interferons, TNF-binding proteins, drugs acting on immunophilins, or antibodies with known impact on the immune system).
* Current treatment or treatment within the past 3 months or planned treatment with drugs known to be toxic to the lens, retina, or the optic nerve.
* Use of any investigational drug or device within 3 months or 5 half-lives of Day 1, whichever is longer, or plans to participate in another study of a drug or device during the trial period.
* Any prior receipt of genetic or stem-cell therapy for ocular or non-ocular disease.

Ages: 0 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular adverse events (AEs) | 24 months
  Incidence and severity of ocular adverse events (AEs)
Incidence and severity of non-ocular adverse events (AEs) | 24 months
  Incidence and severity of non-ocular adverse events (AEs)

SECONDARY OUTCOMES:
Change from baseline to Month 12 in Best-corrected visual acuity (BCVA) | 12 months
  Mean change in BCVA relative to baseline after 12 months of treatment
Change from baseline to Month 12 in retinal sensitivity measured by Full-field stimulus testing (FST) | 12 months
  Mean change in retinal sensitivity measured by FST relative to baseline after 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: ProQR Medical Monitor, Study Director — ProQR Therapeutics
Locations (9):
- Universitair Ziekenhuis Gent (UZ), Ghent, Belgium
- Brazil (2):
  - INRET Clinica e Centro de Pesquisa / Santa Casa BH, Belo Horizonte
  - Federal University of Sao Paulo - Hospital Sao Paulo, São Paulo
- University of Alberta, Edmonton, Alberta, Canada
- Germany (2):
  - Justus-Liebig Universität - Department of Ophthalmology, Giessen
  - University of Tübingen - Institute for Ophthalmic Research, Tübingen
- Eye Clinic University of Campania Liugi Vanvitelli, Naples, Italy
- Amsterdam University Medica Center - Locatie AMC, Amsterdam, Netherlands
- Moorfields Eye Hospital - NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://www.proqr.com